CLINICAL TRIAL: NCT05707754
Title: A Randomized Trial of a Sphenopalatine Ganglion Block With Bupivacaine for Acute Headache
Brief Title: Sphenopalatine Ganglion Block Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-14616
Record Dates: First submitted 2023-01-22; First posted 2023-02-01 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Sphenopalatine Ganglion Nerve Block
Keywords: Sphenopalatine ganglion nerve; Peripheral nerve block; Headache; Migraine
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — Bupivacaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (4):
- High dose with unilateral administration (Active Comparator): High dose (3ml) with unilateral administration of bupivacaine
  Interventions: Drug: Bupivacaine; Device: angiocatheter
- High dose with bilateral administration (Active Comparator): High dose (3ml) with bilateral administration of bupivacaine
  Interventions: Drug: Bupivacaine; Device: angiocatheter
- Low dose with unilateral administration (Active Comparator): Low dose (1ml) with unilateral administration of bupivacaine
  Interventions: Drug: Bupivacaine; Device: angiocatheter
- Low dose with bilateral administration (Active Comparator): Low dose (1ml) with bilateral administration of bupivacaine
  Interventions: Drug: Bupivacaine; Device: angiocatheter

INTERVENTIONS:
Drug: Bupivacaine — Topically applied to sphenopalatine ganglion
Device: angiocatheter — Introduced into nose to reach sphenopalatine ganglion nerve

SUMMARY:
The goal of this clinical trial is to compare the administration and dosage of bupivacaine for sphenopalatine ganglion (SPG) nerve block. The main question[s] it aims to answer are:

* Does a high dose (3ml) give more relief than a low dose (1ml)?
* Does bilateral administration give more relief than unilateral? Participants with headaches will be asked to lie down and have SPG block performed.

Researchers will compare dosage and administration to see how symptoms are reduced.

ELIGIBILITY:
Inclusion Criteria:

* Present to ED for management of headache
* Headache is moderate or severe in intensity

Exclusion Criteria:

* Allergy to bupivacaine
* Nasal or sinus surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Number of participants demonstrating sustained headache relief | 48 hours
  A standard ordinal headache intensity scale will be used for participants to describe their headache as either "severe", "moderate", "mild", or "none". The number of participants who are able to achieve a headache level of "mild" or "none" in the ED within 30 minutes of procedure/medication administration and without requiring additional analgesic medication, and not relapsing to a headache level worse than "mild" during the 48 hours after medication administration, will be determined

SECONDARY OUTCOMES:
Number of participants demonstrating satisfaction with the procedure/medication | 48 hours
  Satisfaction with the procedure/medication as evidenced by the number of participants who provide an affirmative response to the question "Do you want to receive the same procedure/medication the next time you come to the ER with migraine?"

OTHER OUTCOMES:
Number of participants demonstrating improvement in 0-10 pain scale | 60 minutes
  Pain will be assessed using an 11-point numerical rating scale (NRS) as recommended for use in migraine research by the International Headache Society. The NRS scale asks subjects to assign their pain a number between 0 and 10, with 0 = no pain and 10 = worst pain imaginable. Pain scores will be ascertained prior to procedure and at one hour

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Friedman, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No